CLINICAL TRIAL: NCT05456360
Title: Implementation of Digital Vital Sign Monitoring to Decrease Sleep Interruption and Enhance Recovery in Phase II of the PROmoting Sleep, Patient Engagement and Recovery (PROSPER) Project
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor accrual and poor patient engagement with survey completion
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0190; NCI-2022-05712 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention group (Other): Participants will receive sleep enhancement intervention and will wear the ViSi Mobile device.
  Interventions: Device: ViSi Mobile device
- Control group (Other): Participants will receive sleep enhancement intervention only. Participants in the control group will not wear the ViSi Mobile device.
  Interventions: Drug: Sleep enhancement intervention

INTERVENTIONS:
Device: ViSi Mobile device — Participants will wear the device on your wrist like a watch, and it will continuously (non-stop) monitor your pulse, blood pressure, temperature, breathing rate, heart rate, and pulse rate
  Arms: Intervention group
Drug: Sleep enhancement intervention — Participants will receive a medication administration will be limited to before bedtime.
  Arms: Control group

SUMMARY:
This phase II/III trial examines how a sleep enhancement intervention, including the use of wearable digital vital sign monitoring device (ViSi), affects the quality of life of cancer patients receiving acute care. Sleep enchancement interventions may improve the quality of life of patients with cancer due to fewer interruptions at night during hospital stays.

DETAILED DESCRIPTION:
Objective:

Primary Objective:

1). Investigate the impact of our sleep enhancement intervention, that entails a wearable digital vital sign monitoring device, on variation in the quality of life of acute care cancer patients

Secondary Objectives:

1. . Assess the impact of our sleep enhancement intervention on acute care utilization e.g. length of stay, 30-day readmissions
2. . Assess the implementation and feasibility of wearable digital vital signs capture in an inpatient oncologic setting using validated instruments such as system usability scale (SUS) and Weiner implementation outcomes (AIM, FIM, IAM).
3. . Assess the impact, via validated survey instruments, of our sleep enhancement intervention on patient mood, patient activation and satisfaction with inpatient stay experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years of age), english speaking, able to complete consent and survey materials.
* Patients must be admitted to the hospital for at least 3 nights.
* Patient's using pharmacological sleeping aides will be included in the study as this will help us understand if the intervention will also help patients with pre-exisitng sleep disturbances.

Exclusion Criteria:

* Vulnerable populations (pregnancy, incarcerated, history of delirium, suicidal ideation, ischemic stroke with measurable neurologic deficit, cerebral palsy, seizures), primary brain tumor/metastases patients.
* Patients concurrently enrolled in contact isolation with SARS-CoV2 will be excluded.
* Lastly, hospice or hospice-bound patients will also be excluded.
* Any patient can remove themselves from the study at any point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Gottumukkala, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2023 and October 2023, we enrolled 89 patients. 52 patients were assigned to the control group, while 37 were assigned to the intervention group. The study was terminated due to insufficient staff and the inability to enroll an adequate number of patients. Consequently, we could not draw any conclusions.
Groups:
- Standard of Care: Vital Signs were monitor per standard of care
- Intervention: Passive Vital Signs Monitoring: Vital Signs were monitor per PROSPER algorithm
Period: Overall Study
Arm/Group | Standard of Care | Intervention: Passive Vital Signs Monitoring
Started | 52 | 37
Completed | 16 | 9
Not Completed | 36 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Intervention: Passive Vital Signs Monitoring | Total
Number analyzed (Participants) | 52 | 37 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 22 | 56
  >=65 years | 18 | 15 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 10 | 40
  Male | 22 | 27 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 45 | 34 | 79
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 47 | 31 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 37 | 89

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Questionnaires (EuroQol Group EQ-5D)
Description: Score Scales (0-100) 0-worst health/100 best health
Time Frame: through study completion, an average of 1 year
Population: Based on the feedback from the team it was unrealistic to complete the protocol in the estimated period due to lack of patient interest and engagement, data was not collected.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Events were monitored during patients' admission. Admission Time average was 3.5 days
Arm/Group | Standard of Care | Intervention: Passive Vital Signs Monitoring
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/37
Other Adverse Events (participants affected / at risk) | 0/52 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT05456360/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT05456360/ICF_001.pdf